CLINICAL TRIAL: NCT05953948
Title: Intelligent Case Manage Platform to Improve Self-management and Health-related Outcome Among Liver Transplant Recipients: Connection with Artificial Intelligence and Deep Learning
Brief Title: Effectiveness of Intelligent Case Manage Platform in Liver Transplant Recipients
Acronym: ICMP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Weng, Li-Chueh, Professor, Chang Gung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ICMP20230704
Record Dates: First submitted 2023-07-03; First posted 2023-07-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Liver Transplant Disorder; Self Efficacy; Quality of Life
Keywords: liver transplantation; self-efficacy; self-management behavior; health-related quality of life
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: In the feasibility evaluation stage, 200 patients will be recruited for the study. In the quasi-experiment stage, 133 patients will be involved in this experiment: 44 in the experimental group and 89 in the control group. The intervention or usual care will conduct parallel.
Who Masked: Outcomes Assessor
Masking Description: The study participants will be aware they are in the experimental or control group; however, the data collector did not know which group the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intelligent case manage platform (ICMP) and self-management program (Experimental): The experimental group received ICMP information. They could interact with the care manager via chatbot. The ICMP was established with information related to care instruction after liver transplantation.
  Interventions: Other: Intelligent Case Manage Platform (ICMP) and self-management program
- usual care (No Intervention): Participants in the control only received the usual care that included wound care, medication, and infection control.

INTERVENTIONS:
Other: Intelligent Case Manage Platform (ICMP) and self-management program — This platform includes information and instruction related to the care of liver transplantation. Participants could gain knowledge and skill to manage their conditions after liver transplantation.
  Arms: Intelligent case manage platform (ICMP) and self-management program

SUMMARY:
This study is a prospective, quasi-experimental design, with an experimental group and a control group, will be created. The aims of this study are as follows: 1. Describe the self-management and information needs of liver transplant recipients, 2. Create content or modules related to the self-management of liver transplant recipients, 3. Build an intelligent case management platform, 4. Evaluate the usability of the platform, and 5. Conduct deep learning and examine the effects of the intelligent case management platform on self-efficacy, self-management, health outcomes, and health-related quality of life. Data will be collected at discharge (baseline data) and 1, 3, 6, 9, and 12 months after discharge. An estimated 133 patients will be involved in this experiment: 44 in the experimental group and 89 in the control group. Statistical package software (SPSS 22.0) will be used to analyze the data. A generalized estimation equation model will examine the differences in self-efficacy, self-management, and health-related quality of life between the experimental and control groups. Survival analysis and the Kaplan-Meier method will be used to analyze health outcomes, including hospital readmission, emergency visits, episodes of infection and rejection of organs, and death.

DETAILED DESCRIPTION:
Background: Liver transplant recipients require proper self-management to avoid the risk of various complications, reduce hospital readmission and medical costs, and improve their quality of life. They also face diverse challenges in self-management. Therefore, enhancing the self-management of liver transplant recipients after liver transplantation is important. Hospitals and medical facilities taking care of such patients should facilitate individualized care, access to healthcare resources, and planned post-discharge support. The use of information technology, artificial intelligence, and deep learning to identify and confirm the characteristics and types of self-management requirements of liver transplant recipients and provide individualized self-management may help improve their self-management skills and health outcomes. The quality and continuity of care can also be improved. However, no studies have been conducted in this regard.

Purpose: To establish an intelligent case management platform that combines artificial intelligence and deep learning to enhance the self-efficacy and self-management of liver transplant recipients, thereby improving clinical outcomes and health-related quality of life. The aims of this study are as follows: 1. Describe the self-management and information needs of liver transplant recipients, 2. Create content or modules related to self-management of liver transplant recipients, 3. Build an intelligent case management platform, 4. Evaluate the usability of the platform, and 5. Conduct deep learning and examine the effects of the intelligent case management platform on self-efficacy, self-management, health outcomes, and health-related quality of life.

Methods and materials: This study is a prospective, quasi-experimental design, with an experimental group and a control group, will be created. First, the self-management care and information needs of liver transplant patients will be integrated to create the foundation of the intelligent case management platform. For this purpose, an estimated 50 liver transplant recipients and 10 medical staff will be interviewed. The data will be analyzed by qualitative content analysis. Based on these contents, the intelligent case management platform will be developed and evaluated. For the evaluation, data from 200 liver transplant recipients will be collected to assess platform availability, performance, and usage status. Data related to the recipient's use of the platform and reception of self-management from the platform will also be collected for deep learning. The importance and clinical relevance of self-management provided by the platform will be assessed by the medical staff involved in liver transplant care. Deep learning techniques will be utilized, and the effectiveness of the intelligent case management platform in terms of self-efficacy, self-management, health outcomes, and health-related quality of life will be examined. An estimated 133 patients will be involved in this experiment: 44 in the experimental group and 89 in the control group. Data will be collected at discharge (baseline data) and 1, 3, 6, 9, and 12 months after discharge from the hospital. Statistical package software (SPSS 22.0) will be used to analyze the data. A generalized estimation equation model will analyze the differences in self-efficacy, self-management, and health-related quality of life over time between the experimental and control groups. This study proposes innovative applications for information technology, deep learning, and artificial intelligence. It is hoped that multidisciplinary cooperation can improve liver transplant recipients' self-management and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients
* Age 20 years and above
* Ability to use smart-phone

Exclusion Criteria:

* liver encephalopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the score of self-management behavior | Chang of the score from baseline self-management behavior at 1, 3, 6, 9, and 12 months after liver transplantation
  Change of the score of self-management behavior related to the care after liver transplantation assessed by the Self-Management Behavior Scale
Change of the score of self-efficacy | Chang of the score from baseline self-efficacy at 1, 3, 6, 9, and 12 months after liver transplantation
  Change of the score of self-efficacy about manage the condition after liver transplantation assessed by the Self-Efficacy Scale
Change of the score of health-related quality of life | Chang of the score from baseline health-related quality of life at 1, 3, 6, 9, and 12 months after liver transplantation
  Change of the score of health-related quality of life assessed by the questionnaire of Medical Outcome Survey - Short Form 12 (MOS SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chueh Weng, PHD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, TY, Taiwan

IPD SHARING:
Plan to Share IPD: No
We could not share the individual data because of the privacy.